CLINICAL TRIAL: NCT05670730
Title: A Phase 1/2, Randomized, Placebo-controlled, Double-blind, Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamic Effects of Single and Multiple Ascending Doses of AOC 1044 Administered Intravenously to Healthy Adult Volunteers and Participants With DMD Mutations Amenable to Exon 44 Skipping
Brief Title: Study of AOC 1044 in Healthy Adult Volunteers and Participants With Duchenne Muscular Dystrophy (DMD) Mutations Amenable to Exon 44 Skipping
Acronym: EXPLORE44
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Avidity Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AOC 1044-CS1
Record Dates: First submitted 2022-12-06; First posted 2023-01-04 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Duchenne Muscular Dystrophy; Exon 44
Keywords: EXPLORE44; Avidity Biosciences; Avidity; AOC 1044
MeSH Terms: conditions — Muscular Dystrophy, Duchenne | interventions — Sodium Chloride

STUDY DESIGN:
Intervention Model Description: AOC 1044-CS1 (EXPLORE44) is a 2-part study:
  Part A: 5 cohorts with single ascending doses conducted in healthy adult volunteers
  Part B: 3 cohorts with multiple ascending doses in participants with DMD mutations amenable to exon 44 skipping
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- AOC 1044-CS1 Part A - Single Dose Levels 1-5 (Experimental): AOC 1044 will be administered once.
  Interventions: Drug: AOC 1044
- AOC 1044-CS1 Part A - Single Dose: Placebo (Placebo Comparator): Placebo will be administered once.
  Interventions: Drug: Placebo
- AOC 1044-CS1 Part B - Multiple Ascending Dose Levels 1-3 (Experimental): AOC 1044 will be administered three times.
  Interventions: Drug: AOC 1044
- AOC 1044-CS1 Part B - Multiple Ascending Dose: Placebo (Placebo Comparator): Placebo will be administered three times.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AOC 1044 — AOC 1044 will be administered via intravenous (IV) infusion
  Arms: AOC 1044-CS1 Part A - Single Dose Levels 1-5; AOC 1044-CS1 Part B - Multiple Ascending Dose Levels 1-3
Drug: Placebo — Placebo will be administered via intravenous (IV) infusion.
  Other Names: Saline
  Arms: AOC 1044-CS1 Part A - Single Dose: Placebo; AOC 1044-CS1 Part B - Multiple Ascending Dose: Placebo

SUMMARY:
AOC 1044-CS1 (EXPLORE44) is a Phase 1/2 study to evaluate the safety, tolerability, pharmacokinetics, and pharmacodynamic effects of single and multiple ascending doses of AOC 1044 in healthy adult volunteers and participants with DMD mutations amenable to exon 44 skipping.

Part A is a single dose design with multiple cohorts (dose levels) in healthy adult volunteers.

Part B is a multiple-ascending dose design with 3 cohorts (dose levels) in participants with Duchenne.

ELIGIBILITY:
Part A:

Key Inclusion Criteria:

* Aged 18 to 55 years, inclusive, at the time of informed consent
* Body mass index (BMI) of 18.5 to 32.0 kg/m2

Key Exclusion Criteria:

* Clinically significant abnormalities in laboratory results, ECGs, or vitals
* Current or recent use of prescription or nonprescription drugs
* Positive drug/alcohol test at Screening or Day -1
* Elevated blood pressure (BP) >130/80 mmHg at Screening
* Participation in a clinical study in which an investigational product was received within 1 month of screening or 5 half-lives of the investigational product
* Blood or plasma donation within 16 weeks of planned AOC 1044 administration Note: Other protocol defined Inclusion/Exclusion criteria may apply

Part B:

Key Inclusion Criteria:

* Aged 7 to 27 years, inclusive, at the time of informed consent
* Clinical diagnosis of DMD or clear onset of DMD symptoms at or before the age of 6 years
* Confirmation of DMD gene mutation amenable to exon 44 skipping
* Weight ≥ 23 kg
* Ambulatory or non-ambulatory

  * Ambulatory participants: LVEF ≥50% and FVC≥50%
  * Non-ambulatory participants: LVEF ≥45% and FVC≥40%
* PUL 2.0 entry item A ≥3
* If on corticosteroids, stable dose for 30 days before screening and throughout the study

Key Exclusion Criteria:

* Biceps brachii muscles unsuitable for biopsy
* Serum hemoglobin < lower limit of normal
* Uncontrolled hypertension or diabetes
* Prior treatment with any cell or gene therapy
* Prior treatment with another exon 44 skipping agent within 6 months prior to informed consent
* Recently treated with an investigational drug
* History of multiple drug allergies

Ages: 7 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 70 (Actual)
Dates: Start 2022-11-09 (Actual); Primary Completion 2024-11-25 (Actual); Study Completion 2024-11-25 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events (TEAEs) | Through study completion, up to Day 85 (Part A) or Day 169 (Part B)

SECONDARY OUTCOMES:
Plasma pharmacokinetic (PK) parameters | Through Week 8 (Part A); Through Week 12 (Part B)
  Maximum plasma concentration (Cmax) of AOC 1044
Plasma pharmacokinetic (PK) parameters | Through Week 8 (Part A); Through Week 12 (Part B)
  Terminal half-life (T1/2) of AOC 1044
Plasma pharmacokinetic (PK) parameters | Through Week 8 (Part A); Through Week 12 (Part B)
  Area under the concentration-time curve (AUC) of AOC 1044
PMO44 levels in skeletal muscle tissue | Through Week 4 (Part A); Through Week 16 (Part B)
Urine pharmacokinetic parameters | Day 1-2 (0-24 hours after first dose) (Part A); Day 1-2 (0-24 hours after first dose) (Part B)
  Fraction of PMO44 excreted in urine
Change from baseline in exon skipping as measured in skeletal muscle (Part B only) | Baseline, Week 16
Absolute change from baseline in dystrophin protein level in skeletal muscle (Part B only) | Baseline, Week 16
Percentage change from baseline in dystrophin protein level in skeletal muscle (Part B only) | Baseline, Week 16

CONTACTS AND LOCATIONS:
Overall Officials: Carmen Castrillo, MD, Study Director — Avidity Biosciences, Inc.
Locations (10):
- United States (10):
  - Arkansas Children's, Little Rock, Arkansas
  - UCSD, La Jolla, California
  - Stanford University, Palo Alto, California
  - Rare Disease Research - Atlanta, Atlanta, Georgia
  - University of Iowa, Iowa City, Iowa
  - University of Massachusetts Chan Medical School, Worcester, Massachusetts
  - Gillette Children's, Saint Paul, Minnesota
  - Rare Disease Research NC, Hillsborough, North Carolina
  - Abigail Research Institute at Nationwide Children's Hospital, Columbus, Ohio
  - Worldwide Clinical Trials (Part A only), San Antonio, Texas